CLINICAL TRIAL: NCT04045925
Title: Feasibility Study of the Taïso Practice in Parkinson's Disease
Acronym: Taïso-Park
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2019-A01551-56
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Parkinson Disease
Keywords: Taïso; Physical therapy; Exercice therapy; Parkinson disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Taïso practice (Experimental): 6 months of biweekly practice Taïso
  Interventions: Other: Taïso

INTERVENTIONS:
Other: Taïso — Taiso is a physical preparation practice of which the French Judo Federation is a state delegate. It is practiced in most French dojos. During each course, Taiso's practice works the fundamental motor skills (coordination, static and dynamic balance, locomotion and grip), muscle strengthening, target work by simulated attacks-defenses exercises without blows or projections, relaxation and the specific work of knowledge to fall and rise with graduation and progressivity in the intensity and complexity of the exercises as and when practiced.

SUMMARY:
This is a pilot study of descriptive and analytical, prospective feasibility, monocentric, longitudinal with 6 months of bi-weekly practice of Taïso in patients with Parkinson's disease with mild to moderate postural instability.

The intervention is planned over 6 months (25 consecutive weeks) for the whole project of the patient group. Patients are included in the month before the start of the treatment of the intervention. Four standardized evaluation sessions are conducted: a first evaluation during the first week of Taiso and then every 8 weeks (2 months, 4 months and 6 months). Incident collection and fitness assessment tests are performed by the physical trainer while the balance and are performed by a physiotherapist. The quality of life assessment and the MDS-UPDRS II rating are performed during the inclusion visit and then the final study visit (within 2 weeks) after 6 months of practice) with the coordinating neurologist. An evaluation of incidents is also carried out during this end-of-study visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and <85 years old,
* Parkinson's disease diagnosed by a neurologist, treated and sensitive to dopaminergic treatment without limitation of the duration of the disease since the date of diagnosis,
* Patient with mild to moderate postural instability (equivalent to grade 2.5 and 3 on the Hoehn and Yahr scale),
* Naive patient of any practice of Taiso,
* Patient available to perform the Taïso program planned in the study,
* Patient with written informed consent

Exclusion Criteria:

* Patient with a contraindication to the practice of sport
* Pregnant woman, parturient and breastfeeding mother
* Patient deprived of liberty by administrative or judicial decision
* Patient admitted to a health or social facility for purposes other than that of research
* Adults under guardianship or trusteeship or unable to express consent
* Patient not affiliated to a social security system
* Patient already participating in a therapeutic research protocol that aims to improve physical or mental abilities

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Number of traumatic incident(s) and/or cardiovascular(s) | The collection of traumatic and/or cardiovascular incidents will begin in the first Taiso class and continue until the final visit with the neurologist (6 months of collection
  The main judgement criterion is the number of traumatic incident(s) and/or cardiovascular(s) during Taiso practice and on journeys between home and the site of practice until the end of patient participation in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU d'Angers, Angers, France